CLINICAL TRIAL: NCT03621449
Title: Velocity Time Integral vs PICCO for Evaluation of Passive Leg Raising in Septic Shock
Acronym: VIPS
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: RegionSkane ICU 1
Record Dates: First submitted 2018-05-17; First posted 2018-08-08 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Septic Shock
Keywords: passive leg raising; fluid responsiveness; pulse contour analysis; transthoracic ultrasound; velocity time integral
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the present study is to investigate accuracy of changes in cardiac output following passive leg raising as estimated by transthoracic ultrasound as method to predict fluid responsiveness and compare that to changes in cardiac output following PLR as estimated by calibrated pulse contour analysis as method to predict fluid responsiveness in patients with septic shock.

DETAILED DESCRIPTION:
One method to predict fluid responsiveness is to increase preload by transferring blood from the lower extremities to the central compartment through a passive leg raising (PLR) maneuver and then measure the resulting change in cardiac output. It was recently suggested that an increase in cardiac output following PLR had a high accuracy compared other methods to test fluid responsiveness. Different methods to estimate change in cardiac output have been used in studies investigating accuracy of PLR. Most commonly calibrated pulse contour analysis has been used in mechanically ventilated patients whereas transthoracic echocardiography (TTE)has been used in spontaneously breathing patients. While TTE offers the advantage of being less invasive than calibrated pulse contour analysis it is technically challenging and user dependent and the accuracy of the two methods has not been compared.

ELIGIBILITY:
Inclusion Criteria:

1. Septic shock according to the sepsis-3 criteria
2. The treating physician plans to administer fluid to improve organ perfusion and oxygenation due to signs of inadequate organ perfusion and hypoxia (skin mottling, tachycardia (>100), urine output below 0.5 ml/kg/h, lactate persistently > 2 mmol/l and central venous oxygen saturation < 70%, increasing doses of vasoconstrictors to maintain mean arterial pressure >65 mmHg.
3. Hemodynamic monitoring with transpulmonary thermodilution initiated as part of routine clinical monitoring.

Exclusion Criteria:

1. Any condition that will affect the reliability of the PLR procedure or is a contraindication to PLR (compression stockings or intraabdominal pressure > 12 mm Hg, raised intracranial pressure).
2. PaO2/FiO2 < 100 mmHg (13.3 kPa) or suspicion of cardiogenic edema
3. Transthoracic echo does not allow recording of VTI.
4. Age >18 years.
5. No informed consent
6. Prior inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to either of the two study sites a fulfilling inclusion criteria
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operator characteristics curve for prediction of fluid responsiveness. | Cardiac output will be measured immediately prior to passive leg raising and 1 minute after completion of passive leg raising
  Prediction of fluid responsiveness by evaluation change in cardiac output using either transthoracic ultrasound or calibrated pulse contour analysis after a passive leg raising.

SECONDARY OUTCOMES:
Positive and negative likelihood ratios | Cardiac output will be measured immediately prior to passive leg raising and 1 minute after completion of passive leg raising
  Prediction of fluid responsiveness by evaluation change in cardiac output using either transthoracic ultrasound or calibrated pulse contour analysis after a passive leg raising.

OTHER OUTCOMES:
Usefulness | During screening or during examination
  Number of eligible patients in which respective method could not be used

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bentzer, MD, PhD, Principal Investigator — Medical faculty, Lund University
Locations (2):
- Sweden (2):
  - Helsingborg Hospital, Helsingborg
  - Skåne University Hospital, Malmo